CLINICAL TRIAL: NCT05433168
Title: Randomized Cross-over Pilot Study Evaluating the Effectiveness of Shiatsu on Fatigue in Patients With Axial Spondyloarthritis
Brief Title: Study Evaluating the Effectiveness of Shiatsu on Fatigue in Patients With Axial Spondyloarthritis
Acronym: SFASPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CHRO-2021-14
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Spondyloarthritis
Keywords: SHIATSU; axial spondyloarthritis; FATIGUE; CROSS OVER STUDY
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis; Fatigue | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Monocentric randomized controlled cross-over trial with allocation of patients according to a ratio (1:1)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHIATSU GROUP (Experimental): The patients will benefit from shiatsu treatments by a professional according to the shiatsu protocol developed by the Syndicate's evaluation commission Shiatsu Professionals (SPS).
  Interventions: Procedure: SHIATSU; Procedure: DUMMY SHIATSU
- DUMMY SHIATSU GROUP (Experimental): Exercising a fake shiatsu is a real problem as opinions differ. The consensus of the different schools and styles of the technique is that shiatsu pressure is weight transfer. We are therefore going to remove this aspect from the SFASPA shiatsu protocol. The professional will run the same sequence of points, without any weight transfer, being only in contact with the receiver.
  Interventions: Procedure: SHIATSU; Procedure: DUMMY SHIATSU

INTERVENTIONS:
Procedure: SHIATSU — The patients will benefit from shiatsu treatments by a professional according to the shiatsu protocol developed by the Syndicate's evaluation commission Shiatsu Professionals (SPS).
Procedure: DUMMY SHIATSU — Exercising a fake shiatsu is a real problem as opinions differ. The consensus of the different schools and styles of the technique is that shiatsu pressure is weight transfer. We are therefore going to remove this aspect from the SFASPA shiatsu protocol. The professional will run the same sequence of points, without any weight transfer, being only in contact with the receiver

SUMMARY:
Spondyloarthritis is a potentially serious disease with reduced life expectancy. Even if the clinical presentation is eminently variable from one patient to another, the most frequently encountered manifestations such as inflammatory spinal pain, peripheral arthritis or even extra-articular involvement of the disease all represent disabling symptoms, origin of pain, temporary or in some cases permanent functional incapacity, but also general repercussions on daily life (asthenia, reactive depressive syndrome, etc.) which require a multidisciplinary approach, involving several medical, paramedical and other stakeholders, The objective of treatment is to improve quality of life, to control symptoms and inflammation, to prevent structural damage, particularly in peripheral damage, to preserve or restore functional capacities, autonomy and social participation of patients with spondyloarthritis.

In France, the main professional reference for shiatsu is the Syndicat des Professionnels de Shiatsu, which proposes the following definition to define shiatsu:

Shiatsu (finger pressure in Japanese) is an energetic manual discipline addressing the individual as a whole. Shiatsu is part of personal assistance. He receives himself, dressed in soft clothes. Shiatsu is a discipline of well-being and prevention for better health. Its objective is to correct both the energy flow (ki, blood, lymph, etc.) and the body structure (muscles, tendons, etc.) by applying rhythmic pressure to the whole body, most often with the inches. It is for everyone and at all ages. Its principle of action is to restore the free flow of Ki (qi, Energy) in the body.

Shiatsu is a set of pressures performed mainly with the thumbs and the palms of the hands on different areas of the body, often taking up the points of the acupuncture meridians. Shiatsu pressures can be (Ishizuka 1993; Kagotani 1984; Okamoto 2016):

* mobile in a given place and lasting 3 to 5 seconds: a phase of increasing pressure followed by a short holding time then release,
* static: same phases but with a hold time of up to approximately 1 minute or even longer.

To date, there is no treatment specifically targeting fatigue in axSpA. Indeed, the underlying mechanisms of fatigue in SpA remain poorly understood, and could for example involve pro-inflammatory cytokines and the inflammatory process, and/or psychological distress. The effectiveness of non-pharmacological interventions and in particular the care provided by shiatsu practitioners have not been the subject of studies evaluating, according to the criteria of evidence-based medicine, the benefit of this practice, particularly in the context of treatment of spondyloarthritis.

DETAILED DESCRIPTION:
To investigate the variations in the fatigue score (FACIF-F) after a shiatsu intervention (3 sessions) versus a sham shiatsu intervention (3 sessions) (control group).

The primary endpoint will be the percentage of patients responding to the FACIT Fatigue score. A response to fatigue will be defined as an improvement, i.e. an increase of ≥ 4 points in the FACIT-F score corresponding to the minimum clinically important difference.

Monocentric randomized controlled cross-over trial with allocation of patients according to a ratio (1:1) The study will be offered prospectively and systematically to patients with spondyloarthritis meeting the inclusion criteria during a follow-up consultation or in a day hospital or traditional hospitalization in the rheumatology department.

ELIGIBILITY:
Inclusion Criteria:

* The patients with spondyloarthritis meeting the ASAS criteria and followed in the rheumatology department of the Orléans Regional Hospital Center.
* Men and women aged 18 to 70
* Patients with digital or visual analog rating scale ≥ 3 on the 1st question of the BASDAI

Exclusion Criteria:

* Patient with a pathology that contraindicates the practice of shiatsu (evolving infectious skin pathology that would make shiatsu treatment difficult)
* Previous shiatsu treatment
* Inability to attend appointments for the duration of the study
* Pregnant or breastfeeding woman
* Refusal to participate in the study or to sign the consent
* Patients not affiliated or not beneficiaries of a social security scheme
* Person under guardianship or curatorship
* Patient with an uncontrolled epileptic or psychotic condition which, in the opinion of the investigator, would interfere with the smooth running of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients responding to the FACIT Fatigue score | Day 0
  A response to fatigue will be defined as an improvement, i.e. an increase of ≥ 4 points in the FACIT-F score corresponding to the minimum clinically important difference.
  It is a short, easy to administer, 13-item tool that measures a person's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all tired to 0 = very tired)
Percentage of patients responding to the FACIT Fatigue score | Day 14
  A response to fatigue will be defined as an improvement, i.e. an increase of ≥ 4 points in the FACIT-F score corresponding to the minimum clinically important difference.
  It is a short, easy to administer, 13-item tool that measures a person's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all tired to 0 = very tired)
Percentage of patients responding to the FACIT Fatigue score | Day 28
  A response to fatigue will be defined as an improvement, i.e. an increase of ≥ 4 points in the FACIT-F score corresponding to the minimum clinically important difference.
  It is a short, easy to administer, 13-item tool that measures a person's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all tired to 0 = very tired)
Percentage of patients responding to the FACIT Fatigue score | Day 35
  A response to fatigue will be defined as an improvement, i.e. an increase of ≥ 4 points in the FACIT-F score corresponding to the minimum clinically important difference.
  It is a short, easy to administer, 13-item tool that measures a person's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (4 = not at all tired to 0 = very tired)

SECONDARY OUTCOMES:
Global Pain Evaluation (EVN) | Day 0
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 3
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 14
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 18
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 28
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 35
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
Global Pain Evaluation (EVN) | Day 56
  The EVA pain scale is a graduated ruler ranging from 0 to 10. 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 0
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 3
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI Bath Ankylosing Spondylitis Disease Activity Index | Day 14
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 18
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 28
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 35
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit.
BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) | Day 56
  This is a questionnaire to calculate the activity index of ankylosing spondylitis.
  The intensity of 5 symptoms during the past week will be estimated, giving a score from 0 to 10, knowing that 0 means the absence of the symptom and 10 its presence in the highest degree 0 = no pain 10 = maximum imaginable pain Pain will be assessed by the patient at each visit. Show the differences in disease progression between the 2 treatment arms
BASFI questionnaire (Bath ankylosing spondylitis functional index) | Day 0
  It was developed specifically to assess joint mobility in SpA. The BASFI reflects the functional impact, that is to say the inability to perform actions of daily life. For each of the ten activities, you must rate from 0 to 10 the ease or difficulty of performing them during the past month. 0 means completely easy, 10 means impossible. This score is an aid in monitoring ankylosing spondylitis.
  Show the differences in disease progression between the 2 treatment arms
BASFI questionnaire (Bath ankylosing spondylitis functional index) | Day 14
  It was developed specifically to assess joint mobility in SpA. The BASFI reflects the functional impact, that is to say the inability to perform actions of daily life. For each of the ten activities, you must rate from 0 to 10 the ease or difficulty of performing them during the past month. 0 means completely easy, 10 means impossible. This score is an aid in monitoring ankylosing spondylitis.
  Show the differences in disease progression between the 2 treatment arms
BASFI questionnaire (Bath ankylosing spondylitis functional index) | Day 28
  It was developed specifically to assess joint mobility in SpA. The BASFI reflects the functional impact, that is to say the inability to perform actions of daily life. For each of the ten activities, you must rate from 0 to 10 the ease or difficulty of performing them during the past month. 0 means completely easy, 10 means impossible. This score is an aid in monitoring ankylosing spondylitis.
  Show the differences in disease progression between the 2 treatment arms
BASFI questionnaire (Bath ankylosing spondylitis functional index) | Day 35
  It was developed specifically to assess joint mobility in SpA. The BASFI reflects the functional impact, that is to say the inability to perform actions of daily life. For each of the ten activities, you must rate from 0 to 10 the ease or difficulty of performing them during the past month. 0 means completely easy, 10 means impossible. This score is an aid in monitoring ankylosing spondylitis.
  Show the differences in disease progression between the 2 treatment arms
Short Form-36 (SF-36) | Day 0
  It is a self-assessment quality of life scale comprising 11 questions
  Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes:
Short Form-36 | Day 14
  It is a self-assessment quality of life scale comprising 11 questions
  Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes:
Short Form-36 | Day 28
  It is a self-assessment quality of life scale comprising 11 questions.
  Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes:
Short Form-36 | Day 35
  It is a self-assessment quality of life scale comprising 11 questions.
  Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes:
AsQoL Questionnaire (Ankylosing Spondylitis Quality of Life Questionnaire) | Day 0
  Score validated in French in 2010(Pham et al. 2010), it is composed of 18 double-choice (yes/no) items. All the points obtained are added together and divided by the maximum possible total Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes: AS Quality of Life (ASQOL)
AsQoL Questionnaire (Ankylosing Spondylitis Quality of Life Questionnaire) | Day 14
  Score validated in French in 2010(Pham et al. 2010), it is composed of 18 double-choice (yes/no) items. All the points obtained are added together and divided by the maximum possible total Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes: AS Quality of Life (ASQOL)
AsQoL Questionnaire (Ankylosing Spondylitis Quality of Life Questionnaire) | Day 28
  Score validated in French in 2010(Pham et al. 2010), it is composed of 18 double-choice (yes/no) items. All the points obtained are added together and divided by the maximum possible total Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes: AS Quality of Life (ASQOL)
AsQoL Questionnaire (Ankylosing Spondylitis Quality of Life Questionnaire) | Day 35
  Score validated in French in 2010(Pham et al. 2010), it is composed of 18 double-choice (yes/no) items. All the points obtained are added together and divided by the maximum possible total Show the differences in disease progression between the 2 treatment arms for Change in quality of life assessed according to the following indexes: AS Quality of Life (ASQOL)
BASMI measurement index | Day 0
  It allows to evaluate the mobility of the spine. It is composed of 5 items including: cervical rotation, tragus wall distance, lateral flexion of the spine, lumbar flexion and inter malleolar distance. The score for each item is added together to result in a rating out of 10.
BASMI measurement index | Day 35
  It allows to evaluate the mobility of the spine. It is composed of 5 items including: cervical rotation, tragus wall distance, lateral flexion of the spine, lumbar flexion and inter malleolar distance. The score for each item is added together to result in a rating out of 10.
SpA Patient Health Index (ASAS Health Index) | Day 0
  This self-assessment questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EFs) in patients with SpA. The ASAS HI contains items covering the following categories: pain, emotional functions, sleep, sexual functions, mobility, autonomy and community life
SpA Patient Health Index (ASAS Health Index) | Day 14
  This self-assessment questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EFs) in patients with SpA. The ASAS HI contains items covering the following categories: pain, emotional functions, sleep, sexual functions, mobility, autonomy and community life
SpA Patient Health Index (ASAS Health Index) | Day 28
  This self-assessment questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EFs) in patients with SpA. The ASAS HI contains items covering the following categories: pain, emotional functions, sleep, sexual functions, mobility, autonomy and community life
SpA Patient Health Index (ASAS Health Index) | Day 35
  This self-assessment questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EFs) in patients with SpA. The ASAS HI contains items covering the following categories: pain, emotional functions, sleep, sexual functions, mobility, autonomy and community life
Work Productivity Index (WPAI) (Work Productivity and activity Impairment questionnaire) | Day 0
  This is a self-administered questionnaire where the assessment is based on the patient's absenteeism, his presence and his difficulties in carrying out his work or his outside activities. The higher the score, the more the patient has difficulty
Work Productivity Index (WPAI) (Work Productivity and activity Impairment questionnaire) | Day 14
  This is a self-administered questionnaire where the assessment is based on the patient's absenteeism, his presence and his difficulties in carrying out his work or his outside activities. The higher the score, the more the patient has difficulty
Work Productivity Index (WPAI) (Work Productivity and activity Impairment questionnaire) | Day 28
  This is a self-administered questionnaire where the assessment is based on the patient's absenteeism, his presence and his difficulties in carrying out his work or his outside activities. The higher the score, the more the patient has difficulty
Work Productivity Index (WPAI) (Work Productivity and activity Impairment questionnaire) | Day 35
  This is a self-administered questionnaire where the assessment is based on the patient's absenteeism, his presence and his difficulties in carrying out his work or his outside activities. The higher the score, the more the patient has difficulty
Anxiety and Depression (HAD) scale | Day 0
  The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores to be obtained (maximum score for each score = 21)
Anxiety and Depression (HAD) scale | Day 14
  The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores to be obtained (maximum score for each score = 21)
Anxiety and Depression (HAD) scale | Day 28
  The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores to be obtained (maximum score for each score = 21)
Anxiety and Depression (HAD) scale | Day 35
  The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores to be obtained (maximum score for each score = 21)
Pittsburgh Sleep Quality Index (PSQI) | Day 0
  This index is used to assess the sleep quality of subjects over the past month. The 17 scoring items in this study were combined into six components: sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorder, and daytime dysfunction.
  Each component used a Likert4 score (scored from 0 to 3), and the scores were added to obtain a total of 0-21 points. The higher the PSQI index, the worse the quality of sleep. A PSQI >7 is considered indicative of a sleep disorder.
Pittsburgh Sleep Quality Index (PSQI) | Day 14
  This index is used to assess the sleep quality of subjects over the past month. The 17 scoring items in this study were combined into six components: sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorder, and daytime dysfunction.
  Each component used a Likert4 score (scored from 0 to 3), and the scores were added to obtain a total of 0-21 points. The higher the PSQI index, the worse the quality of sleep. A PSQI >7 is considered indicative of a sleep disorder.
Pittsburgh Sleep Quality Index (PSQI) | Day 28
  This index is used to assess the sleep quality of subjects over the past month. The 17 scoring items in this study were combined into six components: sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorder, and daytime dysfunction.
  Each component used a Likert4 score (scored from 0 to 3), and the scores were added to obtain a total of 0-21 points. The higher the PSQI index, the worse the quality of sleep. A PSQI >7 is considered indicative of a sleep disorder.
Pittsburgh Sleep Quality Index (PSQI) | Day 35
  This index is used to assess the sleep quality of subjects over the past month. The 17 scoring items in this study were combined into six components: sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorder, and daytime dysfunction.
  Each component used a Likert4 score (scored from 0 to 3), and the scores were added to obtain a total of 0-21 points. The higher the PSQI index, the worse the quality of sleep. A PSQI >7 is considered indicative of a sleep disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, PH, Principal Investigator — CHR d'Orléans
Locations (1):
- CHU Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernardinelli N, Valery A, Barrault D, Dorland JM, Palut P, Toumi H, Lespessailles E. Effectiveness of Shiatsu on Fatigue in Patients with Axial Spondyloarthritis: Protocol for a Randomized Cross-Over Pilot Study. Rheumatol Ther. 2023 Aug;10(4):1107-1117. doi: 10.1007/s40744-023-00558-w. Epub 2023 May 12. PMID 37173568